CLINICAL TRIAL: NCT04109053
Title: Ultrasensitive Electroanatomic Mapping to Adjudicate Endpoints for Ablation In Paroxysmal AF Patients Using Cryoballoon
Status: Withdrawn | Type: Observational
Why Stopped: PI did not move forward with study
Sponsor: BayCare Health System (Other)
Responsible Party: Sponsor
Other Study IDs: Ultrasensitive EAM
Record Dates: First submitted 2019-09-27; First posted 2019-09-30 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Ultrasensitive Electroanatomic Mapping to Adjudicate Endpoints for Ablation In Paroxysmal AF Patients Using Cryoballoon

DETAILED DESCRIPTION:
Collected data include procedural parameters relevant to pulmonary vein isolation as outlined in the protocol section, DE identified patient demographics, follow up information including rhythm status, antiarrhythmic medication usage, and symptoms or signs to suggest procedural complications relevant to the pulmonary vein isolation procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing pulmonary vein isolation using cryoballoon at St. Joseph's Hospital in FL that sign informed consent

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing pulmonary vein isolation using cryoballoon at St. Joseph's Hospital in FL that sign informed consent
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03-02 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of acute pulmonary vein isolation as adjudicated by pacing catheter based entrance/exit block, and Orion derived activation and voltage map. | 12 months

SECONDARY OUTCOMES:
AT/AF free survival | 12 months
Procedural endpoints including total procedure time, LA dwell time, total flouro time, total ablation time, and total mapping time. | 12 months

IPD SHARING:
Plan to Share IPD: No